CLINICAL TRIAL: NCT00062374
Title: An Evaluation of Preoperative Chemotherapy With Irinotecan and Cisplatin for Advanced, But Resectable Gastric Cancer: A Coordinated Multidisciplinary, Multicenter Study Linking Functional Imaging, Genomic Expression Profiles and Histopathology
Brief Title: Irinotecan and Cisplatin in Treating Patients Who Are Undergoing Surgery For Locally Advanced Cancer of the Stomach or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01438; NCI-2012-01438 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5917; CDR0000304738; MSKCC-03032; 03-032 (Other: Memorial Sloan-Kettering Cancer Center); 5917 (Other: CTEP); P30CA008748 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Gastric Adenocarcinoma; Stage II Gastric Cancer; Stage III Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorodeoxyglucose F18; alovudine; Irinotecan; Magnetic Resonance Spectroscopy

ARMS (1):
- Treatment (preoperative chemotherapy) (Experimental): Neoadjuvant chemotherapy: Patients receive cisplatin IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1, 8, 22, and 29. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Surgery: Within 4 weeks after completion of neoadjuvant chemotherapy, patients undergo radical subtotal or total gastrectomy with lymph node dissection.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Fludeoxyglucose F-18; Other: Fluorothymidine F-18; Drug: Irinotecan Hydrochloride; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo FDG and FLT PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Fludeoxyglucose F-18 — Undergo FDG-PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Fluorothymidine F-18 — Undergo FLT-PET/CT
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; Fluorothymidine F 18
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
Procedure: Positron Emission Tomography — Undergo FDG and FLT PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Therapeutic Conventional Surgery — Undergo radical subtotal or total gastrectomy with lymph node dissection

SUMMARY:
This phase II trial is studying how well giving irinotecan together with cisplatin works in treating patients who are undergoing surgical resection for locally advanced cancer of the stomach or gastroesophageal junction. Drugs used in chemotherapy, such as irinotecan and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug and giving them before surgery may shrink the tumor so that it can be removed during surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the correlation of fluorodeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT) imaging early in the preoperative treatment program of locally advanced gastric cancer with histologic response assessment and patient outcome, defined as overall and progression-free survival.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy and safety of preoperative chemotherapy with irinotecan and cisplatin in the treatment of locally advanced gastric cancer.

II. To examine the biology of locally advanced gastric cancer and the response to chemotherapy by DNA microarray technology and by histopathology.

III. To obtain preliminary data on biodistribution, dosimetry and explore the potential clinical usefulness of fluorodeoxythymidine (FLT) PET in patients with locally advanced gastric cancer undergoing a novel combination neoadjuvant chemotherapy.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Neoadjuvant chemotherapy: Patients receive cisplatin intravenously (IV) over 30 minutes followed by irinotecan IV over 30 minutes on days 1, 8, 22, and 29. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Surgery: Within 4 weeks after completion of neoadjuvant chemotherapy, patients undergo radical subtotal or total gastrectomy with lymph node dissection.

Patients undergo fluorodeoxyglucose FDG-PET/CT at baseline. Some patients undergo additional FDG-PET/CT scans in weeks 3 and 6. Approximately 5 patients undergo fluorothymidine FLT-PET/CT at baseline, during week 3, and/or before surgical resection.

Patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have microscopically confirmed adenocarcinoma of the stomach or gastroesophageal (GE) junction with material reviewed by the Department of Pathology of the participating Institution; tumors involving the GE junction must have the bulk of their disease in the stomach; tumors of the distal esophagus that extend less than 2cm into the stomach are ineligible for this study; using the Siewert's classification for the GE junction, tumors designated as Types II and III are indeed considered eligible for this clinical trial
* All patients must have localized cancer potentially curable by surgery; the tumor stage should be Tany N+ M0 or T3-T4 Nany M0, by staging that includes a computed tomography (CT) scan and either laparoscopy-assisted pancreatobiliary (LAP) or endoscopic ultrasound (EUS); patients with T1-2N0M0 tumors, confirmed by LAP ("good risk") are ineligible; any sites of suspected M1 disease by these criteria must be proven to be M0 prior to entrance into a neoadjuvant trial
* Patients must have a Karnofsky Performance Status >= 60% (Eastern Cooperative Oncology Group [ECOG] =< 2) and be able to tolerate the proposed surgical procedure and chemotherapy regimen
* Patients may not have received prior chemotherapy or radiation for this disease
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000/mm^3
* Serum creatinine =< 1.5 mg/dL
* Total serum bilirubin =< 1.5 mg/dL
* Patients must have signed informed consent indicating that they are aware of the investigational nature of the study and that participation is voluntary
* No clinically significant auditory impairment
* No clinically significant peripheral neuropathy
* New York Heart Association (NYHA) class I-II
* Patients must not have a prior history of cancer within the last five years except for non-melanoma skin cancer, non-metastatic prostate cancer or carcinoma in situ of the uterine cervix

Exclusion Criteria:

* Any metastatic disease
* NYHA Class III or IV heart disease; history of active angina or myocardial infarction within 6 months; history of significant ventricular arrhythmia requiring medication with antiarrhythmics or a history of a clinically significant conduction system abnormality
* Pregnant or lactating women are ineligible; fertile men and women, unless using effective contraception, are ineligible; a pregnancy test will be performed on sexually active women of childbearing potential prior to entry into the study; treatment may not begin until the results of the pregnancy test are ascertained
* Serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy
* Grade 2 or greater pre-existing peripheral neuropathy
* Psychiatric disorders rendering patients incapable of complying with the requirements of the protocol
* Any concurrent active malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer or carcinoma-in-situ of the uterine cervix; patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial
* Clinically significant hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date Opened to Accrual: 6/5/2003 Date Closed to Accrual: 8/8/2006 Date Closed: 6/28/2011 Recruitment location is the medical clinic
Groups:
- Arm I: Cisplatin + Irinotecan
Period: Overall Study
Arm/Group | Arm I
Started | 55
Completed | 43
Not Completed | 12
Not completed — Not treated | 12

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Neoadjuvant chemotherapy: Patients receive cisplatin IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1, 8, 22, and 29. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Surgery: Within 4 weeks after completion of neoadjuvant chemotherapy, patients undergo radical subtotal or total gastrectomy with lymph node dissection.
  irinotecan hydrochloride: Given IV
  cisplatin: Given IV
  conventional surgery: Undergo radical subtotal or total gastrectomy with lymph node dissection
  positron emission tomography/computed tomography: Undergo FDG-PET/CT
  fludeoxyglucose F 18: Undergo FDG-PET/CT
  positron emission tomography/computed tomography: Undergo FLT-PET/CT
  fluorine F 18 fluorothymidine: Undergo FLT-PET/CT
Arm/Group | Arm I
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Histological Response Determined by FDG Uptake Correlates
Description: The primary objective was to demonstrate that a decrease in FDG-SUV discriminates treatment response. Response was defined pathologically based on microscopic inspection for residual cancer cells and fibrosis.
  Using a two sample t-test, we would be able to adequately test that the decrease in SUV early in the treatment plan is significantly different between responders and non responders. Data adjudication was invalid, and needs to be re-adjudicated
  Non-Responder= Tumor Regression Grade 3 or higher Responder=Tumor Regression Grade 1 (CR) or Grade 2 (PR)
Time Frame: Day 15
Population: Technical problems with measurement of FDG-SUV data leading to unreliable or uninterpretable data. Data adjudication was invalid, and needs to be re-adjudicated. Therefore, only histological response is reported.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 43
participants
  Progression of Disease | 2
  Responders | 3
  Non-Responders | 38

2. Other Pre Specified Outcome: Disease Free Survival (DFS)
Description: Overall Survival (OS) and Disease Free Survival (DFS) are the secondary endpoints. Technical problems with measurement of OS leading to unreliable or uniterpretable data. Data adjudication was invalid, and needs to be re-adjudicated. Therefore, only DFS data is being reported.
Time Frame: Every 3 mos for the first 2 yrs, then every 6 mos for 2 years and once a year afterwards, up to 5 years
Population: Technical problems with measurement leading to unreliable or uninterpretable data. Data adjudication was invalid, and needs to be re-adjudicated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 43
months | 23.8 [14 to NA] — The value is infinity.

ADVERSE EVENTS:
Description: Number of participants at risk is the same as the total number of participants that were treated.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 14/55
Other Adverse Events (participants affected / at risk) | 44/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=55)
Abdominal pain/cramping (Gastrointestinal disorders) | 1 (1)
CNS/cerebrovascular ischemia (Nervous system disorders) | 2 (2)
Cardiovascular, other (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Hemorrhage, NOS (Blood and lymphatic system disorders) | 2 (3)
Hemoglobin decrease (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=55)
Abdominal pain/cramping (Gastrointestinal disorders) | 15 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 16 (18)
Constipation (Gastrointestinal disorders) | 4 (5)
Creatinine (Investigations) | 6 (43)
Dehydration (Metabolism and nutrition disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 25 (41)
Dizziness (Nervous system disorders) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Edema (General disorders) | 6 (6)
Fatigue (General disorders) | 36 (83)
Hemoglobin decrease (Blood and lymphatic system disorders) | 30 (54)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (20)
Hyperkalemia (Metabolism and nutrition disorders) | 11 (12)
Hypernatremia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 35 (219)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 16 (31)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (41)
Hyponatremia (Metabolism and nutrition disorders) | 20 (60)
Hypophosphatemia (Metabolism and nutrition disorders) | 17 (31)
Hearing impaired (Ear and labyrinth disorders) | 4 (4)
White blood cell count decrease (Investigations) | 32 (148)
Lymphocyte count decrease (Investigations) | 11 (37)
Mood alteration/anxiety (Psychiatric disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 33 (64)
Neuropathy-sensory (Nervous system disorders) | 11 (12)
Neutrophil count decrease (Investigations) | 31 (112)
Pain, other (General disorders) | 3 (3)
Platelet count decreased (Investigations) | 21 (81)
Aspartate aminotransferase increase (Investigations) | 7 (14)
Alanine aminotransferase increase (Investigations) | 10 (31)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Taste disturbance (Nervous system disorders) | 4 (6)
Thrombosis (Vascular disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 12 (23)
Weight loss (Investigations) | 5 (6)

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to unreliable or uninterpretable data. Data adjudication was invalid, and needs to be re-adjudicated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less